CLINICAL TRIAL: NCT06238427
Title: Impact of Timing of Soft Tissue Augmentation to Increase Width of Keratinized Mucosa Around Dental Implant
Brief Title: Soft Tissue Augmentation Around Dental Implant
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: A11100221
Record Dates: First submitted 2023-12-28; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2023-12

CONDITIONS: Gingival Atrophy
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Group 1 participants underwent free gingival graft placement two months before implant placement.
- Group2: Group 2 in which the participants underwent the placement of the free gingival graft during the second stage of surgery, specifically at the time of healing abutment placement

SUMMARY:
Patients were randomly distributed into two groups (G1 and G2), all patients were treated by a submerged dental implant protocol and free gingival graft (FGG) harvested from the palate as follows:

* Group 1 (G1), received the FGG two months before implant placement.
* Group 2 (G2), received the FGG at the time of second-stage surgery (i.e. at the time of healing abutment placement).

All periodontal and radiographic assessments were done by the same operator who was neither involved in the evaluation nor the distribution process. The operator did all the evaluation steps and was completely blinded to the treatment protocol.

DETAILED DESCRIPTION:
In this investigation, a randomized clinical trial was employed. The patient's randomization was completed by one of the department's senior residents, who was not involved in the trial and was unaware of any relevant treatment plan. A computer-generated randomization list used a randomization table to perform the randomization (SPSS v23.0). Patients were randomly distributed into two groups (G1 and G2), all patients were treated by a submerged dental implant protocol and FGG harvested from the palate. All patients received a thorough description of all procedures involved in the study. Signing a written consent was mandatory for being enrolled in the study. Complete medical and dental histories were recorded for all patients and complete clinical intraoral and extraoral examinations were done for all patients.

Selected patients were questioned about the cause and time of extractions, whether extractions were because of periodontal disease, dental decay or other causes. Previous experiences with dental procedures were also discussed. Intraoral photographs were taken to record the existing condition of teeth and mucosa before implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 years or older
* Systemic Condition: Healthy
* Keratinized Mucosa Width: Less than 2mm at the intended implant site
* Bucco-lingual Bone Width: At least 5.5 mm in a single edentulous space
* Mesio-distal Distance: At least 7 mm between adjacent teeth in a single edentulous space
* Minimal Bone Height: Not less than 10 mm
* Residual Alveolar Ridge: Healthy and well-formed, covered with firm mucosa
* Periodontal Health: Absence of signs of periodontal bone loss or significant soft tissue .loss in teeth adjacent to the implant site
* Inter-arch Space: Adequate, exceeding 7 mm

Exclusion Criteria:

* Cooperation: Uncooperative patients
* Pregnancy: Individuals with known pregnancies
* Parafunctional Habits: Abnormal parafunctional habits such as bruxism and clenching
* Systemic Illnesses: Patients with systemic illnesses that could disrupt healing
* Medication: Individuals receiving systemic corticosteroids or other drugs impacting .osseointegration or post-operative healing
* Smoking: Smokers consuming more than 10 cigarettes per day

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty patients (12 female / 8 male) seeking dental implant placement due to missing teeth and deficient keratinized mucosa width were enrolled in this observational study. The study population was selected from patients attending the clinic of the Periodontology Department of Oral Medicine and Periodontology at Mansoura University. Recruitment occurred from July 2019 to June 2022..
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Keratinized Mucosa Width (KMW) | Baseline, 1 month, 3 months, 6 months, and 9 months
  Measurement Method: The assessment of KMW involved measuring from the alveolar ridge zenith to the muco-gingival junction (MGJ) using a calibrated periodontal probe.
  Unit of Measure: Millimeters (mm)
Soft Tissue Thickness (STT) | Baseline, 1 month, 3 months, 6 months, and 9 months
  Measurement Method: STT was determined 1.5 mm apical to the soft tissue margin (STM) using a short anesthesia needle or endodontic micro-opener with a silicon stopper.
  Unit of Measure: Millimeters (mm) Measurement Procedure: The needle was inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until a hard surface was felt. The silicon stopper was placed in tight contact with the soft tissue surface, and the penetrated part was measured on an endodontic ruler. Measurements were rounded to the nearest half of a millimeter.
Graft Shrinkage | 1 month, 3 months, 6 months, and 9 months
  The decrease in the size of the graft at each follow-up time was compared to the baseline. size. It was presented in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Samah Elmeadawy, Ph.D, Study Director — Mansoura University
Locations (1):
- Wafaa saleh, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No